CLINICAL TRIAL: NCT05585801
Title: Continuous Glucose Monitoring in Intensive Care Unit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Barbora Hagerf, Principal Investigator, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGM 001
Record Dates: First submitted 2022-10-12; First posted 2022-10-19 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Blood Glucose; Critical Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Device: Dexcom G6 continuous glucose monitor
- Control Group (Active Comparator)
  Interventions: Diagnostic Test: Blood glucose measurements according to standards of care

INTERVENTIONS:
Device: Dexcom G6 continuous glucose monitor — Continuous glucose monitor will be used to measure interstitial glucose and aid in guiding the insulin therapy to achieve target blood glucose range of 6-10 mmol/l.
  In the control group, blood glucose will be measured according to standards of care and a blinded continuous monitor will be used to compare the time i range between the arms.
  Arms: Intervention Group
Diagnostic Test: Blood glucose measurements according to standards of care — Blood glucose will be measured using point of care glucose meter and standard biochemistry methods. Blinded CGM will be applied to obtain continuous glucose values for post-hoc comparison.
  Arms: Control Group

SUMMARY:
Glucose control in ICU patients is challenging and exerts high burden on the nursing staff. Continuous glucose monitors (CGM) are now approved and widely available in the outpatient setting for patients with diabetes mellitus. However, only minimal evidence on CGM performance, reliability and benefit in achieving desired glucose control in the intensive care setting has been gathered so far.

The objective of this study is to assess whether the use of CGM helps to maintain blood glucose levels within the time in range recommended for patients in the intensive care.

In addition, accuracy of the sensor will be evaluated and compared to measurements of blood glucose by standardized biochemistry methods.

DETAILED DESCRIPTION:
This will be a non-commercial, investigator-driven, active comparator-controlled, randomized, open-label and non-inferiority clinical study to be performed at the Institute for Clinical and Experimental Medicine in Prague. Patients that are being prepared for one of the surgical procedures mentioned below will be asked to participate:

1. pancreas surgery - total or partial pancreas resection
2. orthotopic liver transplantation
3. simultaneous pancreas and kidney transplantation
4. patients with diabetes mellitus undergoing major surgery

After obtaining the informed consent, they will be randomized into one of two treatment groups:

1. Study arm with continuous glucose monitor added to standard treatment, where the values obtained by CGM will aid in adjusting the insulin treatment.
2. Control arm with blinded continuous glucose monitor that will be treated according to the standard of care, where the CGM data will be collected in a blind fashion and evaluated after completion of the follow-up.

Each surgical group will be randomized and evaluated separately and independently.

Continuous glucose monitoring will be initiated after completing the surgical procedure in order to avoid interferences during the procedure.

Insulin therapy will be adjusted according to the standard in-house ICU protocol for insulin dose adjustment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, of 18 to 80 years of age, undergoing one of the following surgical procedures and post-operative care at ICU:

   1. pancreas surgery - total or partial pancreas resection
   2. orthotopic liver transplantation
   3. simultaneous pancreas and kidney transplantation
   4. patients with diabetes mellitus undergoing major surgery
2. Patient must have signed the Patient Informed Consent Form.

Exclusion Criteria:

Any criteria that would disable surgical procedures involved

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time in target range of 6-10 mmol/l | From the time of continuous glucose sensor insertion, which will be performed after admission to postoperative ICU, until the discharge from postoperative ICU, approx. 5-7 days

SECONDARY OUTCOMES:
Mean blood glucose levels | From the time of continuous glucose sensor insertion, which will be performed after admission to postoperative ICU, until the discharge from postoperative ICU, approx. 5-7 days
Time spent in hyperglycaemia level 1 (glucose levels 10.1-13.9 mmol/l ) | From the time of continuous glucose sensor insertion, which will be performed after admission to postoperative ICU, until the discharge from postoperative ICU, approx. 5-7 days
  Amount of time (%) spent in hyperglycaemia level 1 (glucose levels 10.1-13.9 mmol/l )
Time spent in hyperglycaemia level 2 (glucose levels above 13.9 mmol/l ) | From the time of continuous glucose sensor insertion, which will be performed after admission to postoperative ICU, until the discharge from postoperative ICU, approx. 5-7 days
  Amount of time (%) spent in hyperglycaemia level 2 (glucose levels above 13.9 mmol/l )
Time spent in hypoglycaemia level 1 (glucose levels 3.0-3.8 mmol/l ) | From the time of continuous glucose sensor insertion, which will be performed after admission to postoperative ICU, until the discharge from postoperative ICU, approx. 5-7 days
  Amount of time (%) spent in hypoglycaemia level 1 (glucose levels 3.0-3.8 mmol/l )
Time spent in hypoglycaemia level 2 (glucose levels below 3 mmol/l ) | From the time of continuous glucose sensor insertion, which will be performed after admission to postoperative ICU, until the discharge from postoperative ICU, approx. 5-7 days
  Amount of time (%) spent in hypoglycaemia level 2 (glucose levels below 3 mmol/l )
Glycaemic variability assessed by standard deviation of blood glucose levels | From the time of continuous glucose sensor insertion, which will be performed after admission to postoperative ICU, until the discharge from postoperative ICU, approx. 5-7 days
Glycaemic variability assessed by coefficient of variation (%CV) | From the time of continuous glucose sensor insertion, which will be performed after admission to postoperative ICU, until the discharge from postoperative ICU, approx. 5-7 days
Daily dose of insulin | From admission until the discharge from postoperative ICU, approx. 5-7 days
  Daily dose of insulin and dosing speed throughout the day
Surgical complications | From admission to postoperative ICU until the discharge from hospital, approx. 10-15 days
  Surgical site infections, wound dehiscence, wound leakage
Infectious complications | From admission to postoperative ICU until the discharge from hospital, approx. 10-15 days
  Pneumonia, abdominal sepsis, urosepsis
Time until discharge from the inpatient care | From admission to postoperative ICU until the discharge from hospital, approx. 10-15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Clinical and Experimental Medicine, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Study protocol will be available upon request throughout the study duration. Source data will be available upon request after completion of the study and publication of the results

REFERENCES:
- [Derived] Protus M, Voglova Hagerf B, Jabor A, Franekova J, Nemetova L, Uchytilova E, Indrova V, Beckova J, Macek A, Doleckova M, Svirlochova V, Mraz M, Haluzik M, Girman P, Viravova M, Kohn MA, Klonoff DC, Kieslichova E. Accuracy and feasibility of real-time continuous glucose monitoring in early postoperative intensive care after liver transplantation. Ther Adv Endocrinol Metab. 2026 Jan 9;17:20420188251405372. doi: 10.1177/20420188251405372. eCollection 2026. PMID 41523586